CLINICAL TRIAL: NCT06925711
Title: Investigation of the Effect of Hypotensive Anesthesia on Cognitive Functions in Orthognathic Surgery
Brief Title: The Effect of Hypotensive Anesthesia on Cognitive Functions in Orthognatic Surgery
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Tumay Uludag Yanaral, Associate Professor, Medipol University
Other Study IDs: MEDIPOLU-6143
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Dysfunction; Postoperative Complications
Keywords: orthognathic surgery; hypotensive anesthesia; cerebral oxygen saturation
MeSH Terms: conditions — Cognitive Dysfunction; Postoperative Complications | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients aged 18 years and older with ASA I-II scores who were diagnosed with dentofacial deformity
  Interventions: Device: Near-Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near-Infrared Spectroscopy (NIRS) — Controlled hypotensive anesthesia during orthognathic surgery with cerebral oxygen saturation monitoring using Near-Infrared Spectroscopy (NIRS). NIRS was used to continuously monitor regional cerebral oxygen saturation (rSO2) throughout the procedure to observe the effects of controlled hypotension on cerebral perfusion

SUMMARY:
The purpose of this study is to evaluate the effects of maintaining adequate cerebral oxygen saturation on patients undergoing orthognathic surgery. Orthognathic surgery is performed to repair anomalies in the maxillofacial skeleton for both aesthetic and functional purposes. During these procedures, controlled hypotensive anesthesia is commonly used to reduce bleeding, improve surgical field visibility, and shorten operation time.

In controlled hypotensive anesthesia, mean arterial blood pressure is deliberately reduced to approximately 55-60 mmHg. While this technique offers surgical advantages, it may potentially reduce cerebral blood flow and oxygen saturation, which could affect cognitive function.

This study will investigate the relationship between cerebral oxygen saturation levels maintained during orthognathic surgery and postoperative neuropsychological outcomes. Patients will undergo cognitive assessments before and after surgery while cerebral oxygen saturation is continuously monitored during the procedure. Our findings will help establish safety parameters for hypotensive anesthesia in orthognathic surgery and potentially contribute to improved anesthesia management protocols that better preserve cognitive function.

DETAILED DESCRIPTION:
Orthognathic surgery is a surgical procedure performed to repair anomalies in the maxillofacial skeleton. It can be performed for maxillofacial aesthetics as well as for functional purposes. Since orthognathic surgery is performed in a field where vascular structures are dense, complications such as intraoperative bleeding are likely to occur.

Le Fort I osteotomy and bilateral sagittal split ramus osteotomy (BSSRO) are frequently used treatment methods for dentofacial deformities. Significant bleeding may occur especially during Le Fort I osteotomy. Therefore, controlled hypotensive anesthesia is frequently used during maxillofacial surgery procedures to reduce bleeding, increase the visibility of the surgical field, and prevent blood loss.

During controlled hypotensive anesthesia, mean arterial blood pressure (MAP) is reduced to around 55-60 mmHg. This technique makes the operation more comfortable for both the surgical team and the anesthesia team. Vasoactive and anesthetic agents such as direct-acting vasodilators, autonomic ganglion blockers, beta-adrenergic receptor blockers, and calcium channel blockers are used to provide hypotensive anesthesia.

However, prolonged hypotension may lead to organ damage due to hypoperfusion. Uncontrolled prolongation of systemic hypotension may cause cerebral ischemia, neuronal death, and permanent brain damage by causing a decrease in cerebral blood flow. Cerebral circulation has a complex and unpredictable autoregulatory mechanism. Therefore, it is difficult to maintain the balance between hypotension and cerebral perfusion.

Changes in cerebral blood flow and cerebral tissue perfusion may cause cognitive changes because they affect the nutrition of neural tissues. The aim of this study is to evaluate the effects of controlled hypotensive anesthesia applied in orthognathic surgery on intraoperative cerebral blood flow-cerebral oxygen saturation and cognitive functions of patients and to determine the degree of these effects.

As part of the study, cognitive function tests will be performed on the patient population before and after surgery, and cerebral oxygen saturation will be continuously monitored during surgery. The results may help determine the safety limits of hypotensive anesthesia applied during orthognathic surgery and potentially develop cerebral protection strategies.

The results of this research are expected to contribute to the development of new approaches to improve anesthesia management in patients undergoing orthognathic surgery. Additionally, by testing the hypothesis that maintaining cerebral oxygen saturation may improve cognitive outcomes, it can contribute to increasing patient safety in maxillofacial surgical practices.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing Orthognathic surgery under general anesthesia ASA grade ≤ grade III; Patients can communicate normally, can cooperate and complete cognitive function test; Patients volunteered and signed informed consent.

Exclusion Criteria:

BMI < 18 or > 27 kg / m2; Previous history of dementia, psychosis or other central nervous system diseases or mental diseases, such as cerebral infarction, stroke, Parkinson's disease, etc; Patients taking sedatives or antidepressants; Alcoholics or drug addicts; Patients with cognitive impairment before operation (MMSE score < 23); Patients with peripheral vascular diseases and contraindication of arterial puncture and catheterization; Patients unable to carry out long-term follow-up or poor compliance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of both genders, over 18 years of age, undergoing elective Orthognathic surgery in general anesthesia.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function measured by Mini-Mental State Examination (MMSE) scores | Baseline (7 days before surgery), postoperative 10th day, 1st month, and 3rd month after surgery
  The Mini-Mental State Examination (MMSE) is a 30-point questionnaire used extensively in clinical and research settings to measure cognitive impairment. It will be used to assess changes in cognitive function that may be associated with cerebral oxygen saturation levels during controlled hypotensive anesthesia in orthognathic surgery.

SECONDARY OUTCOMES:
Incidence and severity of cerebral oxygen desaturation events during controlled hypotensive anesthesia | Intraoperatively, from induction of anesthesia until extubation
  Cerebral oxygen saturation (rSO2) will be continuously monitored bilaterally using Near-Infrared Spectroscopy (NIRS) during surgery. Cerebral oxygen desaturation events are defined as a decrease in rSO2 of >20% from baseline or an absolute value <50% lasting more than 15 seconds. The number, duration, and severity of these events will be recorded and analyzed for correlation with cognitive outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Zheng Y, Zhang J. Cerebral oxygenation and hemodynamic changes during ephedrine and phenylephrine administration for transient intraoperative hypotension in patients undergoing major abdominal surgery: a randomized controlled trial. BMC Anesthesiol. 2025 Feb 20;25(1):87. doi: 10.1186/s12871-025-02944-z. PMID 39979813
- [Background] Hsiao YC, Chang YT, Cheng CS, Lien KH. Dexmedetomidine infusion on blood loss in orthognathic surgery: A retrospective study on its efficacy. J Formos Med Assoc. 2025 Feb 13:S0929-6646(25)00051-8. doi: 10.1016/j.jfma.2025.02.009. Online ahead of print. No abstract available. PMID 39952888
- [Background] Ravelo V, Olate S, Bravo-Soto G, Zaror C, Mommaerts M. Systematic review of soft-to-hard tissue ratios in orthognathic surgery: 3D analysis-update of scientific evidence. Int J Oral Maxillofac Surg. 2025 Sep;54(9):819-829. doi: 10.1016/j.ijom.2025.02.008. Epub 2025 Mar 17. PMID 40102081